CLINICAL TRIAL: NCT03630172
Title: The Effect of Dry Needling at the Thoracolumbar Junction on Measures of Sympathetic Outflow and Local and Remote Muscular Flexibility in Subjects With Low Back Pain and Decreased Hamstring Length
Brief Title: Dry Needling at the Thoracolumbar Junction on Measures of Sympathetic Outflow and Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-289-Non-NSU Health
Record Dates: First submitted 2018-07-20; First posted 2018-08-14 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Low Back Pain
Keywords: low back pain; dry needling; flexibility; sympathetic nervous system
MeSH Terms: conditions — Low Back Pain | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to one of two dry needling conditions: dry needling or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Random assignment will occur using opaque envelopes. The primary investigator (who is also the care provider) will select an envelope when a subject arrives. The research assistant, who will be blinded to group allocation, will take the pre and post intervention measurements. The primary investigator will be blinded to the pre and post intervention measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): Dry needles will be sterile, and 0.30 x 60mm in gauge and length. Needles will be placed using an inferomedial approach with the subject positioned in prone. The needle is inserted perpendicular to the skin and then is guided inferiorly and medially until it reaches the lamina. Needles will be manipulated in a "pistoning" fashion for 15 seconds.
  Interventions: Procedure: Dry needling
- Sham Needling Group (Sham Comparator): Non-penetrating needles were constructed by cutting 100mm needles where the handle meets the shaft, and sanding down any rough edges. Guide tubes from 40mm needles will be used. These needles will be place in the same location and manipulated in the same fashion as in the dry needling group, except the needles will not have penetrated the skin.
  Interventions: Procedure: Dry needling

INTERVENTIONS:
Procedure: Dry needling — Using a thin, filiform needle to penetrate a muscle and its trigger point to produce a local twitch response

SUMMARY:
Dry needling (DN) is becoming more frequently performed by physical therapists around the world to treat musculoskeletal pain. Dry needling is a form of trigger point therapy that evolved from using injections of local anesthetics. Although dry needling is becoming more commonly used, there is little agreement on how it works. Researchers have focused their efforts investigating other forms of manual therapy until very recently. To date, no studies have looked at how dry needling effects muscles distant from the area being treated. Most of the body's sympathetic nervous system (fight or flight response) is located in the thoracic spine, it may be a "silent" contributor to musculoskeletal problems in the arms and legs. The purpose of this study is to determine how dry needling the thoracolumbar junction affects pain, flexibility, and other non-invasive measures of nervous system output in people who have low back pain and tightness of their hamstring muscles. Standard dry needling treatment will be compared with a placebo. The investigators hypothesize that dry needling will have a greater sympathetic nervous system response, as measured by changes in heart rate, skin temperature and skin conductance, when compared with the placebo. The investigators also hypothesize that dry needling will have a greater positive effect on flexibility of the low back and hamstring muscles when compared to the placebo.

DETAILED DESCRIPTION:
Although DN is being used more often in treatment of musculoskeletal disorders, there continues to be little agreement about the pathways on which it works. Research on the neurophysiological effects of DN has increased in the past 10 years, however much about the treatment is still poorly understood. A better understanding of the neurophysiological mechanisms on which DN acts, and how it influences structures distant from the site of treatment, can lead to improved choices of therapeutic activities, and potentially superior outcomes.

Many studies have investigated the effects of joint mobilization or manipulation on the sympathetic nervous system (SNS), but fewer studies have investigated the effects of DN. Of the studies on joint mobilization, a large percentage examined treatment to the cervical spine, specifically C5, and tested SNS-related outcomes in the cervical spine, upper thoracic spine, and upper extremities (UEs). The sympathetic nerve fibers that supply the lower extremities (LEs) originate from T10-L2, and future research should investigate the effects on the LE when its direct sympathetic connection is treated.

At this time, there is minimal research on manual therapy treatment to the thoracolumbar (TL) spine and its effect on the LEs. The thoracic spine is the origin of nearly all SNS outflow to the extremities, and should therefore not be overlooked as a potentially "silent" contributor to musculoskeletal dysfunction in the extremities.

The goals of this study are:

1. To quantify the magnitude of the SNS response to DN at the TL junction in subjects with low back pain and decreased hamstring length, using valid measures of SNS activity.
2. To describe the effect of DN at the TL junction on muscle length both local and remote to the site of treatment.
3. To determine if DN to the TL junction has a significantly greater segmental sympatho-excitatory effect than extrasegmental effect, as measured by pressure-pain threshold (PPT) in the LE and UE.
4. To determine if immediate changes in SNS activity after DN are related to clinically meaningful outcomes at 24-hour follow-up.

Research questions for this study are:

1. What are the differences in indicators of SNS activity, such as heart rate variability (HRV), electrodermal activity (EDA), skin temperature (ST) and PPT of the LE, when DN or sham DN is performed at the TL junction in subjects with low back pain and decreased hamstring length?
2. How does DN to the TL junction affect lumbar paraspinal muscle and hamstring length in subjects with low back pain and decreased hamstring length?
3. How far superiorly does the sympatho-excitatory response ascend when DN is performed at the TL junction in subjects with low back pain and decreased hamstring length?
4. Do immediate changes in SNS activity correlate with greater clinical improvements at short-term follow-up, as measured by pain rating, global rating of change (GRC), and the Oswestry Disability Index (ODI)?

Hypotheses for this study are:

H1: DN will cause a greater SNS response than sham DN, as measured by HRV, ST, EDA, and PPT in the LE.

H2: Subjects who receive DN to the TL junction will have a greater improvement in fingertip-to-floor (FTF) measurement, straight leg raise (SLR) and knee extension (KE) measurements from baseline than subjects who receive sham DN.

H3: DN to the TL junction will create a greater sympatho-excitatory effect in the LE when compared with the UE, as measured by PPT.

H4: There is a relationship between immediate changes in sympathetic outflow, as measured by low frequency (LF) to high frequency (HF) ratio of HRV immediately following DN or sham DN, and GRC, ODI, and pain at 24-hour follow-up.

A research proposal has been reviewed and approved by the Institutional Review Board (IRB) of Nova Southeastern University. Subjects will be recruited via advertisements placed in outpatient physical therapy clinics throughout Montgomery and Frederick Counties, in Maryland. A power analysis was performed a priori using G Power (Version 3.1.9.3). Sample size calculation was based on the primary outcome of SNS activity, and PPT was chosen as the primary endpoint because there is the most available data pertaining to PPT after DN treatment. Based on the findings for ipsilateral changes in PPT by Salom-Moreno et al when compared with a control group, 27 subjects in each group (total 54 subjects) will be required to detect an effect size of 0.8 in PPT between the two groups with an alpha level of .05 at a power of 0.8. Subjects will be accepted consecutively and data collection will continue until the desired number of subjects has been reached.

Upon arrival at the clinic, the research assistant will confirm that one limb has greater than or equal to 15o of hamstring restriction at R1 and R2. If both limbs meet the criteria for participation, the most restricted limb will be used for analysis. Subjects will complete a Participant Data Form, Informed Consent with assistance from the primary investigator as needed, the Numeric Pain Rating Scale (NPRS), and the ODI. The NPRS is frequently used scale for quantifying pain. The NPRS is an 11-point scale with anchors of "no pain" and "worst pain imaginable." The ODI is one of the most commonly used disability scales for patients with low back pain. It has been found as a favorable measure for symptoms ranging from mild to severe.20 Excellent test-retest reliability has been proven at 24-hour (r=0.99) and 4-day (r=0.91) follow-ups, and test-retest reliability decreases as the length of time before follow-up increases.

Subjects will be randomly assigned to the treatment group or the sham needling group. Randomization will occur using a simple method of opaque envelopes sealed with index cards indicating the allocated group inside of it. When a subject arrives and is completing the initial paper work, an envelope will be selected and opened by the primary researcher. The research assistant will be blinded to each subject's group, and will take all baseline measurements. These measurements will include PPT, FTF test, KE, and SLR.

PPT will be measured by a Wagner digital algometer (Wagner Instruments, Greenwich, CT, USA) and will be measured in kilograms. Each subject will be instructed to say "stop" when the pressure becomes "slightly unpleasant pain." The maximum pressure at the time the subject says "stop" will be recorded. The mean of three trials will be recorded.

The FTF test assesses total trunk flexion mobility and will be performed in the same manner as Perret et al in their validity and reliability study. A subject will stand without shoes on a 20 cm platform with feet together. While keeping knees, arms, and fingers fully extended, the subject will bend forward as far as possible and the vertical distance between the tip of the middle finger and the platform will be recorded. The FTF test has been shown to have excellent intrarater reliability (ICC=.99). The mean of 3 trials will be used for analysis.

Baseline® digital inclinometers will be used to measure KE and SLR. SLR will be measured in supine with the knee fully extended and the ankle in a resting position. The inclinometer will be placed at the midpoint between the tibial tuberosity and the distal end of the tibia and secured with a Velcro strap. The subjects will be instructed to keep the contralateral limb in contact with the treatment table at all times. The contralateral limb and pelvis will not be stabilized, as research has shown that stabilization does not affect SLR reliability measures. The examiner will record the number of degrees excursion until the first resistance is felt (R1), and then the number of degrees at maximum, pain-free elevation (R2). The mean of three trials will be recorded.

KE will be measured in supine similar to Mason et al in their 2016 study. One inclinometer will be used to maintain 90o hip flexion, while a second inclinometer will be anchored at the midpoint between the tibial tuberosity and the distal end of the tibia. Both will be secured with Velcro straps. The subject's lower leg will be passively extended until the first resistance is felt (R1) and then at the maximum number of degrees of pain-free knee extension (R2).

After all baseline measurements are completed, subjects will be connected to a BIOPAC® data acquisition unit, which will monitor HRV, ST, and EDA. HRV refers to changes in heart rate as well as interbeat intervals, and will be used in this study to determine changes in heart rate secondary to autonomic nervous system (ANS) activation. HRV will be measured by the peak-to-peak intervals when using photoplethysmography (PPG).

ST is a measure of cutaneous circulation, which is mediated by the sympathetic vasoconstrictor and vasodilator nerves. SNS stimulation leads to superficial vasoconstriction, which would lead to a decrease in ST. A ST thermistor transducer will be taped to the dorsal aspect of the foot of the LE that has the greatest hamstring restriction, which will be determine in the baseline testing. Skin thermistor measurements show excellent test-retest reliability, with the typical error <0.1 degree Celcius.

EDA refers to changes in skin conductance when the ANS is stimulated and the sweat glands become more active. They are most concentrated in the palms and plantar surfaces of the feet, so these would be ideal locations for EDA data collection. It is a sensitive and easy method to measure sympathetic arousal, and it is arguably one of the best measures of sympathetic arousal because it does not receive input from the parasympathetic nervous system (PNS). Electrodes with isotonic gel will be placed on the LE that has the greatest hamstring restriction. The active electrode will be on the plantar surface of the foot and the ground electrode will be placed on the dorsal surface of the foot.

An 8-minute acclimation period will occur followed by a 5-minute baseline recording. The primary investigator will perform the treatment condition that was randomly assigned. Proper clean technique will be followed for all subjects, including the subjects receiving the placebo. This will decrease the likelihood that the subject will know which treatment he/she is receiving. The PT administering treatment will wear gloves, and 70% isopropyl alcohol will be used to prepare the skin over the muscles to be treated.

Subjects will be treated on the right and left sides at both segments. All materials will be handled according to Occupational Safety and Health Administration Blood Borne Pathogens standards. Subjects will continue to have SNS output monitored for 5 minutes after treatment has been completed. After the 5-minute period, subjects will be disconnected from the equipment, and the research assistant will complete all follow-up measurements in the exact manner stated earlier in this chapter.

All subjects will attend one follow-up visit approximately 24 hours after their initial visit. The research assistant will gather measurements of FTF, KE, SLR, and PPT of the UE and LE. Subjects will also complete an ODI and a GRC during this visit. GRC is a simple and convenient scale that is used in research and in the clinic to quantify a summation of a patient's improvements in pain, disability, and quality of life. Subjects will be reconnected to the BIOPAC® MP36R data acquisition unit as previously described. They will undergo an 8-minute acclimation period followed by a 5-minute data collection period. The same limb will be monitored as in the subject's initial visit. After data collection is complete, subjects in the sham DN group will be offered DN in the same manner as the DN group.

For H1 two-way ANCOVAs will be used for each dependent variable of SNS activity. Covariates will include pre-intervention measurement scores and level of needle anxiety. For H2 flexibility measurements will be separated into "local" and "remote" tests. The FTF test will quantify local flexibility, and the SLR and KE tests will quantify remote flexibility. A two-way ANCOVA will be use for analysis of local flexibility. The covariate will be the pre-intervention scores. For the remote flexibility analysis, a two-way MANCOVA will be used. The covariate will be the pre-intervention measurements. Post-hoc testing will be performed for H1 and H2 to determine between which factors differences occurred, if applicable. For H3 the data will be analyzed using a t test. Change scores in PPT in the LE will be compared to change scores in the UE, and only the DN group will be included. Prior to conducting the tests, data will be analyzed to be sure they meet the assumptions for each statistical test. For H4 a Pearson's r will be used to determine if there is a statistically significant relationship between SNS output immediately after receiving the treatment condition and the outcomes measures of GRC, change in ODI, and change in NPRS. 17 A 2-point change has been found to be the minimum clinically important difference in patients with low back pain and shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Low Back Pain
2. decreased flexibility greater than or equal to 15 degrees of at least one hamstring, as measured by KE
3. Age 18-70 years

Exclusion Criteria:

1. Local skin lesion, local or systemic infection
2. Previous treatment of DN to any body part
3. History of abnormal bleeding
4. Presence of radicular symptoms
5. Prescription anticoagulant therapy
6. Autoimmune disease, central nervous system disorder, or diabetes
7. Previous surgery to lumbar spine
8. Inability to read and understand English, or cognitive impairment that would limit the ability to give consent.
9. Pregnancy
10. BMI greater than 30 kg/m2

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2019-08-10 (Actual)

PRIMARY OUTCOMES:
Pressure pain threshold | immediately before dry needling or sham condition
  measured via Wagner algometer in kg/cm^2 in upper and lower extremity
Pressure pain threshold | immediately following dry needling or sham condition
  measured via Wagner algometer in kg/cm^2 in upper and lower extremity
Pressure pain threshold | 24 hours after dry needling or sham condition
  measured via Wagner algometer in kg/cm^2 in upper and lower extremity

SECONDARY OUTCOMES:
Oswestry Disability Index | immediately before dry needling or sham condition
  a 10-item questionnaire relating to functional restrictions from back pain
Oswestry Disability Index | 24 hours after dry needling or sham condition
  a 10-item questionnaire relating to functional restrictions from back pain
Numeric Pain Rating Scale | immediately before dry needling or sham condition
  rates current pain level from 0-10
Numeric Pain Rating Scale | immediately after dry needling or sham condition
  rates current pain level from 0-10
Numeric Pain Rating Scale | 24 hours after dry needling or sham condition
  rates current pain level from 0-10
Global Rating of Change | 24 hours after dry needling or sham condition
  an 11-point scale relating to changes in pain, function, and quality of life
Straight Leg Raise | immediately before dry needling or sham condition
  Measured in degrees via digital inclinometry
Straight Leg Raise | immediately after dry needling or sham condition
  Measured in degrees via digital inclinometry
Straight Leg Raise | 24 hours after dry needling or sham condition
  Measured in degrees via digital inclinometry
Knee Extension | immediately before dry needling or sham condition
  Measured in degrees via digital inclinometry
Knee Extension | immediately after dry needling or sham condition
  Measured in degrees via digital inclinometry
Knee Extension | 24 hours after dry needling or sham condition
  Measured in degrees via digital inclinometry
Fingertip to Floor | immediately before dry needling or sham condition
  measured in centimeters from or beyond raised platform
Fingertip to Floor | immediately after dry needling or sham condition
  measured in centimeters from or beyond raised platform
Fingertip to Floor | 24 hours after dry needling or sham condition
  measured in centimeters from or beyond raised platform
Electrodermal Activity | immediately before dry needling or sham condition
  tonic activity of SNS measured via electrodes placed on dorsal and plantar surfaces of the foot
Electrodermal Activity | immediately after dry needling or sham condition
  tonic activity of SNS measured via electrodes placed on dorsal and plantar surfaces of the foot
Electrodermal Activity | 24 hours after dry needling or sham condition
  tonic activity of SNS measured via electrodes placed on dorsal and plantar surfaces of the foot
Skin Temperature | immediately before dry needling or sham condition
  measure via thermistor placed on the dorsum of the foot, measured in degrees Celcius
Skin Temperature | immediately after dry needling or sham condition
  measure via thermistor placed on the dorsum of the foot, measured in degrees Celcius
Skin Temperature | 24 hours after dry needling or sham condition
  measure via thermistor placed on the dorsum of the foot, measured in degrees Celcius
Heart Rate Variability | immediately before dry needling or sham condition
  measured via photoplethysmography; refers to changes in heart rate after sympathetic nervous system stimulation
Heart Rate Variability | immediately after dry needling or sham condition
  measured via photoplethysmography; refers to changes in heart rate after sympathetic nervous system stimulation
Heart Rate Variability | 24 hours after dry needling or sham condition
  measured via photoplethysmography; refers to changes in heart rate after sympathetic nervous system stimulation

CONTACTS AND LOCATIONS:
Overall Officials: Nicole G Clark, MSPT, Principal Investigator — Nova Southeastern University
Locations (1):
- Sports and Orthopaedic Therapy Services, LLC, Kensington, Maryland, United States

REFERENCES:
- [Background] Kingston L, Claydon L, Tumilty S. The effects of spinal mobilizations on the sympathetic nervous system: a systematic review. Man Ther. 2014 Aug;19(4):281-7. doi: 10.1016/j.math.2014.04.004. Epub 2014 Apr 13. PMID 24814903
- [Background] Vicenzino B, Cartwright T, Collins D, Wright A. Cardiovascular and respiratory changes produced by lateral glide mobilization of the cervical spine. Man Ther. 1998;3(2):67-71.
- [Background] Jowsey P, Perry J. Sympathetic nervous system effects in the hands following a grade III postero-anterior rotatory mobilisation technique applied to T4: a randomised, placebo-controlled trial. Man Ther. 2010 Jun;15(3):248-53. doi: 10.1016/j.math.2009.12.008. Epub 2010 Jan 25. PMID 20093065
- [Background] McGuiness J, Vicenzino B, Wright A. Influence of a cervical mobilization technique on respiratory and cardiovascular function. Man Ther. 1997 Nov;2(4):216-220. doi: 10.1054/math.1997.0302. PMID 11440535
- [Background] Chiu TW, Wright A. To compare the effects of different rates of application of a cervical mobilisation technique on sympathetic outflow to the upper limb in normal subjects. Man Ther. 1996 Sep;1(4):198-203. doi: 10.1054/math.1996.0269. PMID 11440508
- [Background] Perry J, Green A. An investigation into the effects of a unilaterally applied lumbar mobilisation technique on peripheral sympathetic nervous system activity in the lower limbs. Man Ther. 2008 Dec;13(6):492-9. doi: 10.1016/j.math.2007.05.015. Epub 2007 Jul 20. PMID 17643340
- [Background] Sterling M, Jull G, Wright A. Cervical mobilisation: concurrent effects on pain, sympathetic nervous system activity and motor activity. Man Ther. 2001 May;6(2):72-81. doi: 10.1054/math.2000.0378. PMID 11414776
- [Background] Schmid A, Brunner F, Wright A, Bachmann LM. Paradigm shift in manual therapy? Evidence for a central nervous system component in the response to passive cervical joint mobilisation. Man Ther. 2008 Oct;13(5):387-96. doi: 10.1016/j.math.2007.12.007. Epub 2008 Mar 3. PMID 18316238
- [Background] Sampath KK, Botnmark E, Mani R, Cotter JD, Katare R, Munasinghe PE, Tumilty S. Neuroendocrine Response Following a Thoracic Spinal Manipulation in Healthy Men. J Orthop Sports Phys Ther. 2017 Sep;47(9):617-627. doi: 10.2519/jospt.2017.7348. Epub 2017 Jul 13. PMID 28704625
- [Background] Abbaszadeh-Amirdehi M, Ansari NN, Naghdi S, Olyaei G, Nourbakhsh MR. Neurophysiological and clinical effects of dry needling in patients with upper trapezius myofascial trigger points. J Bodyw Mov Ther. 2017 Jan;21(1):48-52. doi: 10.1016/j.jbmt.2016.04.014. Epub 2016 Apr 14. PMID 28167189
- [Background] Ozden AV, Alptekin HK, Esmaeilzadeh S, Cihan C, Aki S, Aksoy C, Oncu J. Evaluation of the Sympathetic Skin Response to the Dry Needling Treatment in Female Myofascial Pain Syndrome Patients. J Clin Med Res. 2016 Jul;8(7):513-8. doi: 10.14740/jocmr2589w. Epub 2016 May 29. PMID 27298659
- [Background] Ziaeifar M, Arab AM, Karimi N, Nourbakhsh MR. The effect of dry needling on pain, pressure pain threshold and disability in patients with a myofascial trigger point in the upper trapezius muscle. J Bodyw Mov Ther. 2014 Apr;18(2):298-305. doi: 10.1016/j.jbmt.2013.11.004. Epub 2013 Nov 9. PMID 24725800
- [Background] Ga H, Choi JH, Park CH, Yoon HJ. Dry needling of trigger points with and without paraspinal needling in myofascial pain syndromes in elderly patients. J Altern Complement Med. 2007 Jul-Aug;13(6):617-24. doi: 10.1089/acm.2006.6371. PMID 17718644
- [Background] Gifford L, Thacker M. A clinical overview of the autonomic nervous system, the supply to the gut and mind-body pathways. In: Gifford L, ed. Topical Issues in Pain 3. Bloomington, IN: AuthorHouse UK Ltd; 2013:21-52.
- [Background] Heneghan NR, Rushton A. Understanding why the thoracic region is the 'Cinderella' region of the spine. Man Ther. 2016 Feb;21:274-6. doi: 10.1016/j.math.2015.06.010. Epub 2015 Jul 9. PMID 26189592
- [Background] Salom-Moreno J, Sanchez-Mila Z, Ortega-Santiago R, Palacios-Cena M, Truyol-Dominguez S, Fernandez-de-las-Penas C. Changes in spasticity, widespread pressure pain sensitivity, and baropodometry after the application of dry needling in patients who have had a stroke: a randomized controlled trial. J Manipulative Physiol Ther. 2014 Oct;37(8):569-79. doi: 10.1016/j.jmpt.2014.06.003. Epub 2014 Sep 8. PMID 25199825
- [Background] Williamson A, Hoggart B. Pain: a review of three commonly used pain rating scales. J Clin Nurs. 2005 Aug;14(7):798-804. doi: 10.1111/j.1365-2702.2005.01121.x. PMID 16000093
- [Background] Fritz JM, Irrgang JJ. A comparison of a modified Oswestry Low Back Pain Disability Questionnaire and the Quebec Back Pain Disability Scale. Phys Ther. 2001 Feb;81(2):776-88. doi: 10.1093/ptj/81.2.776. PMID 11175676
- [Background] Jette DU, Halbert J, Iverson C, Miceli E, Shah P. Use of standardized outcome measures in physical therapist practice: perceptions and applications. Phys Ther. 2009 Feb;89(2):125-35. doi: 10.2522/ptj.20080234. Epub 2008 Dec 12. PMID 19074618
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Background] Perret C, Poiraudeau S, Fermanian J, Colau MM, Benhamou MA, Revel M. Validity, reliability, and responsiveness of the fingertip-to-floor test. Arch Phys Med Rehabil. 2001 Nov;82(11):1566-70. doi: 10.1053/apmr.2001.26064. PMID 11689977
- [Background] Atamaz F, Ozcaldiran B, Ozdedeli S, Capaci K, Durmaz B. Interobserver and intraobserver reliability in lower-limb flexibility measurements. J Sports Med Phys Fitness. 2011 Dec;51(4):689-94. PMID 22212274
- [Background] Huguenin L, Brukner PD, McCrory P, Smith P, Wajswelner H, Bennell K. Effect of dry needling of gluteal muscles on straight leg raise: a randomised, placebo controlled, double blind trial. Br J Sports Med. 2005 Feb;39(2):84-90. doi: 10.1136/bjsm.2003.009431. PMID 15665203
- [Background] Mason JS, Crowell M, Dolbeer J, Morris J, Terry A, Koppenhaver S, Goss DL. THE EFFECTIVENESS OF DRY NEEDLING AND STRETCHING VS. STRETCHING ALONE ON HAMSTRING FLEXIBILITY IN PATIENTS WITH KNEE PAIN: A RANDOMIZED CONTROLLED TRIAL. Int J Sports Phys Ther. 2016 Oct;11(5):672-683. PMID 27757280
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Smith AD, Crabtree DR, Bilzon JL, Walsh NP. The validity of wireless iButtons and thermistors for human skin temperature measurement. Physiol Meas. 2010 Jan;31(1):95-114. doi: 10.1088/0967-3334/31/1/007. Epub 2009 Nov 26. PMID 19940348
- [Background] Critchley HD. Electrodermal responses: what happens in the brain. Neuroscientist. 2002 Apr;8(2):132-42. doi: 10.1177/107385840200800209. PMID 11954558
- [Background] Dawson M, Schell AM, Filion DL. The Electrodermal System. Handbook of Psychophysiology: Cambridge University Press; 2000:200-223
- [Background] Braithwaite JJ, Watson DG, Jones R, Rowe M. A guide for analysing electrodermal activity (EDA) and skin conductance responses (SCRs) for psychological experiments. University of Birmingham, UK: Behavioral Brain Sciences Centre; 2013
- [Background] Tuvblad C, Isen J, Baker LA, Raine A, Lozano DI, Jacobson KC. The genetic and environmental etiology of sympathetic and parasympathetic activity in children. Behav Genet. 2010 Jul;40(4):452-66. doi: 10.1007/s10519-010-9346-0. Epub 2010 Feb 17. PMID 20162348
- [Background] Freeman R, Chapleau MW. Testing the autonomic nervous system. Handb Clin Neurol. 2013;115:115-36. doi: 10.1016/B978-0-444-52902-2.00007-2. PMID 23931777
- [Background] Bloodborne pathogens. Occupational Safety and Health Standards, Z, Toxic and Hazardous Substances. Washington, DC: United States Department of Labor Occupational Safety and Health Administration.
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. Spine (Phila Pa 1976). 2005 Jun 1;30(11):1331-4. doi: 10.1097/01.brs.0000164099.92112.29. PMID 15928561
- [Background] Michener LA, Snyder AR, Leggin BG. Responsiveness of the numeric pain rating scale in patients with shoulder pain and the effect of surgical status. J Sport Rehabil. 2011 Feb;20(1):115-28. doi: 10.1123/jsr.20.1.115. PMID 21411827